CLINICAL TRIAL: NCT02179996
Title: Comparison of Two Vaccinal Schemes for DTP-Pertussis-Hib Primo-immunisation in Very Preterm-born Neonates: a Randomised Bicentric Controlled Study
Brief Title: Diphtheria, Tetanus, Poliomyelitis -Pertussis-Hib Immunisation in Preterm-born Neonates
Acronym: VacciPrema
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Rachel VIEUX, Professor Rachel Vieux, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-A01377-28
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Hib Immunisation in Very Preterm-born Infants; Pertussis Immunisation in Very Preterm-born Infants
Keywords: Vaccination; Very preterm-born infants; Hib immunisation; Pertussis immunisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Three vaccine injections (Active Comparator): Infants in this study arm will receive three vaccine injections at two, three and four months after birth (vaccine: DTP-pertussis-Hib).
  Interventions: Biological: Three vaccine injections DTP-pertussis-Hib
- Two vaccine injections (Experimental): Infants in this study arm will receive two vaccine injections at two and four months after birth (vaccine: DTP-pertussis-Hib).
  Interventions: Biological: Two vaccine injections DTP-pertussis-Hib

INTERVENTIONS:
Biological: Three vaccine injections DTP-pertussis-Hib — DTP-pertussis-Hib injections at two, three, four months after birth
  Arms: Three vaccine injections
Biological: Two vaccine injections DTP-pertussis-Hib — DTP-pertussis-Hib injections are administered at two and four months after birth
  Arms: Two vaccine injections

SUMMARY:
Preterm neonates are fragile to infections. Their immune system is immature, yet in France, primary vaccines are injected at two months of age, as in term infants.

Recommendations for vaccinations in infants have changed in France in 2013, suppressing the second injection at three months after birth. Preterm and full-term born infants are now vaccinated at two and four months of age, but no data regarding efficacy in very preterm infants have been registered.

The investigators hypothesize that two vaccine injections (at two and four months) would be less efficient than three injections (two, three and four months) in very preterm-born infants.

ELIGIBILITY:
Inclusion Criteria:

* infants born < 33 weeks gestation in Nancy and Thionville Maternity Wards
* signed parental consent

Exclusion Criteria:

* immunodeficiency
* vaccine contra-indication

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Hib antibody dosage in blood sample | 5 months after birth

SECONDARY OUTCOMES:
Pertussis antibody dosage in blood sample | 5 months after birth

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Regional et Universitaire, Maternite Regionale, Nancy
  - Centre Hospitalier de Thionville, Thionville